CLINICAL TRIAL: NCT01561092
Title: Efficacy of Escitalopram Treatment in Acute Stroke and the Role of SERT Genotype in Stroke
Brief Title: Escitalopram Treatment In Acute Stroke
Acronym: ESTIAS
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study medication could not be supplied. An alternative project will be conducted
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 397-2011
Record Dates: First submitted 2012-03-20; First posted 2012-03-22 (Estimated); Last update posted 2012-06-19 (Estimated); Status verified 2012-06

CONDITIONS: Stroke
Keywords: Stroke; RCT; SSRI; Outcome
MeSH Terms: conditions — Stroke | interventions — Escitalopram; Dexetimide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Escitalopram (Active Comparator)
  Interventions: Drug: Escitalopram
- Non active drug (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Escitalopram — 5 or 10 mg escitalopram tablets administered orally once daily
  Other Names: SSRI; Cipralex
  Arms: Escitalopram
Drug: Placebo — Tablets
  Arms: Non active drug

SUMMARY:
Growing international scientific evidence has indicated a positive effect of SSRI treatment (serotonin reuptake inhibitors) after stroke, beyond its antidepressant effect. We wish to conduct a prospective randomised double blind placebo-controlled multicenter study of the combined neuroprotective and antithrombotic effects of SSRI treatment after stroke. Deletion of the SERT (serotonin transporter) gene may influence this treatment effect and may in itself be a risk factor for stroke, an aspect we also wish to explore.

Hypotheses:

1. SSRI treatment commenced in the acute phase of stroke (day 2-5) protects against new thromboembolic events and leads to better rehabilitation.
2. A specific SERT genotype is associated with an increased risk of first ever stroke.
3. A specific SERT genotype is associated with a higher risk of post stroke depression.

600 stroke patients will be randomised to either escitalopram or placebo treatment in a 1:1 ratio and genotyped according to SERT polymorphisms. The treatment and follow up period is 6 months. During these 6 months there will be 2 clinical follow up visits, one telephone control and one visit to evaluate compliance regarding medication. Patients who had an MRI as a part of the routine investigations done upon admission (approximately 300 patients) will have a control MRI after 6 months.

Additionally 400 patients, not eligible for participation i the randomised controlled trial, will be genotyped and answer questionnaires after 1 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* First ever ischemic stroke
* Age 18 years or above

Exclusion Criteria

* Hemorrhagic stroke
* Dementia or other neurodegenerative disease
* Antidepressant treatment within 6 months of admission
* Acute need for antidepressant treatment
* Drug abuse or other conditions that may indicate noncompliant behavior
* Liver failure (increased liver enzyme levels up to or more than 2 times upper limit)
* Renal failure (GFR under 30)
* Hyponatremia (S-potassium below 130 mmol/l)
* Actively bleeding ulcer
* Fatal stroke or other severe co morbidity that markedly decreases expected life span
* Prolonged QT interval (QTc above 500 ms)
* Ongoing treatment with drugs known to prolong the QT interval

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
New vascular events | 6 months

SECONDARY OUTCOMES:
Death of any cause | 6 months
Myocardial Infarction | 6 months
Re-stroke | 6 months
Motor function | 6 months
  Fugl-Meyer Motor score is performed
White Matter lesions | 6 months
  Evaluated on MRI
Bleeding complications | 6 months
Combined vascular death | 6 months
Cognitive abilities | 6 months
  SDMT and MMSE tests are performed

CONTACTS AND LOCATIONS:
Overall Officials: Grethe Andersen, Prof. DMSc, Principal Investigator — University Hospital of Aarhus, Neurology Dept.
Locations (3):
- Denmark (3):
  - Neurology Department, Aalborg Hospital, Aalborg
  - Neurology Department, University Hospital of Aarhus, Aarhus
  - Neurology Department, Glostrup Hospital, Glostrup Municipality